CLINICAL TRIAL: NCT02737865
Title: "The Fingerprint: Spoke-wheel Sign" of Focal Nodular Hyperplasia: Assessment of Novel Ultrasound Approach Using Superb Microvascular Imaging Technique
Brief Title: Superb Microvascular Imaging in Focal Nodular Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Woo Kyoung Jeong, MD, Associate professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-10-134-003
Record Dates: First submitted 2016-01-15; First posted 2016-04-14 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Focal Nodular Hyperplasia
Keywords: Focal nodular hyperplasia; Ultrasonography; Superb-Microvascular imaging; Contrast-enhanced ultrasonography
MeSH Terms: conditions — Focal Nodular Hyperplasia | interventions — Sonazoid; perfluorobutane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMI and sonazoid (single arm) (Experimental): Patients with focal nodular hyperplasia will undergo ultrasonography with Superb-Microvascular imaging and additional sonazoid-enhanced ultrasonography. SMI is a software function in a Toshiba Aplio 500 system. Sonazoid is contrast-material for US and it is a intervention for patient with FNH. Sonazoid will be administered at a dose of 0.015 mL/kg by manual bolus injection, followed by a 10 mL normal saline flush via a peripheral venous line
  Interventions: Drug: Sonazoid; Device: Superb-Microvascular imaging

INTERVENTIONS:
Drug: Sonazoid — Sonazoid: Commercially available contrast material for ultrasonography
  Other Names: Perfluorobutane
Device: Superb-Microvascular imaging — Superb-Microvascular imaging: new sonographic software technique on ultrasonography to detect low-vascular flow without use of contrast media for ultrasonography

SUMMARY:
Focal nodular hyperplasia (FNH) in liver is the second common benign hepatic tumor. It usually shows hypervascular mass on imaging studies and it is not easy to differentiate with other hypervascular malignant tumor. For diagnosis of FNH, contrast-enhanced ultrasonography (US) has been used to detect 'spoke-wheel sign', which can be typically seen in FNH. However, temporal window of vascular phase using contrast-enhanced US (CEUS) is very short (about 10 sec) and coordination of patient's respiration during US exam is absolutely needed. Thus, the investigators will use Superb-Microvascular imaging (SMI, Toshiba, Japan) for detection of 'spoke-wheel sign' in patients with proven FNH, which enable to detect slow micro vascular flow without using CEUS.

First, to compare the detection rate of 'spoke-wheel sign' between CEUS using sonazoid (Perfluorobutane, GE healthcare) and SMI.

Second, to compare the accuracy of size measurement between gray-scale US and SMI (reference standard: CEUS using sonazoid.)

DETAILED DESCRIPTION:
1. To evaluate the detection rate of 'spoke-wheel sign' on CEUS using sonazoid and SMI (primary outcome).

   Each US findings during exam for patients with FNH were recorded by radiologist. The results were interpreted by consensus using 4 scale bar.

   0. Absence of 'spoke-wheel sign'
   1. Mild suspicious of 'spoke-wheel sign'
   2. Highly suspicious of 'spoke-wheel sign'
   3. Definite "spoke-wheel sign'
2. To evaluated the accuracy of size measurement for FNH on gray-scale US and SMI (reference standard: CEUS using sonazoid).

   To calculate the measurement error between each method and CEUS using sonazoid on US images using measurement of maximum diameter of tumor.
3. Sample size calculation according to the primary outcome.

Expecting the detection rate of "spoke-wheel sign" on SMI, 20% (known detection rate on CEUS using sonazoid, 23.5%), a sample size of 62 patients was required using 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy or imaging proven focal nodular hyperplasia

Exclusion Criteria:

1. Pregnant women
2. Patient's age > 70
3. Egg allergy
4. Breast-feeding women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05; Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Grading of spoke-wheel sign on CEUS using sonazoid and SMI in patients with focal nodular hyperplasia | 1 day
  a.To evaluate the detection rate of 'spoke-wheel sign' on CEUS using sonazoid and SMI (primary outcome).
  Each US findings during exam for patients with FNH were recorded by radiologist. The results were interpreted by consensus using 4 scale bar.
  0. Absence of 'spoke-wheel sign'
  1. Mild suspicious of 'spoke-wheel sign'
  2. Highly suspicious of 'spoke-wheel sign'
  3. Definite "spoke-wheel sign'

SECONDARY OUTCOMES:
Measurement error of focal nodular hyperplasia between b-mode US and SMI according to the reference standard, CEUS | 1 day
  To calculate the measurement error between b-mode US and SMI using measurement of maximum diameter of tumor. Reference standard is the size of tumor on sonazoid enhanced US.

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyoung Woo, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Undecided